CLINICAL TRIAL: NCT04838743
Title: A Non-interventional, Single-arm, Multicentre, Prospective Study Investigating the Glycaemic Control and Treatment Pattern Associated With the Use of Xultophy® (IDegLira) in a Real-world Adult Population With Type 2 Diabetes Mellitus in Japan. GOAL (Glycaemic Outcome Assessment IDegLira) Study
Brief Title: GOAL: A Research Study Looking at Long Term Blood Sugar Control in People With Type 2 Diabetes Treated With Xultophy® in Local Clinical Practice in Japan.
Acronym: GOAL
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN9068-4743; U1111-1253-2025 (Other: World Health Organization (WHO)); jRCT1051210008 (Registry Identifier: JAPIC (Japan))
Record Dates: First submitted 2021-04-07; First posted 2021-04-09 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — IDegLira

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IDegLira: Real-world adult population with type 2 diabetes mellitus in Japan.
  Interventions: Drug: IDegLira

INTERVENTIONS:
Drug: IDegLira — Patients will be treated with commercially available Xultophy® (IDegLira) in a pre-filled pen injector (FlexTouch®) at the discretion of the treating physician in accordance with the Xultophy® label in Japan.
  The decision to initiate treatment with Xultophy® is at the treating physician's discretion according to the approved Xultophy® label in Japan and independent from the decision to include the patient in the study.

SUMMARY:
The purpose of this study is to collect information on how Xultophy® works with other oral anti diabetic medication in patients with type 2 diabetes.

Participants will get Xultophy® as prescribed by the study doctor. The study will last for about 26 weeks. Participants will be asked questions about health and diabetes treatment and lab tests as part of normal doctor's appointment.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
* The decision to initiate treatment with commercially available Xultophy® has been made by the patient/Legally Acceptable Representative (LAR) and the treating physician before and independently from the decision to include the patient in this study.
* Male or female, age above or equal to 20 years at the time of signing informed consent
* Diagnosed with T2DM (Type 2 diabetes mellitus ) above or equal to 180 days prior to initiation of Xultophy® treatment.
* Treated with any oral anti-hyperglycaemic medication(s), except for oral GLP-1 RAs, for at least 60 days prior to initiation of Xultophy® treatment.
* Available and documented HbA1c value less or equal to 12 weeks prior to initiation of Xultophy® treatment.

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having given informed consent in this study.
* Participation in any clinical trial of an approved or non-approved investigational medicinal product within 30 days before prior to initiation of Xultophy® (Simultaneous participation in a trial with the primary objective of evaluating an approved or non-approved investigational medicinal product for prevention or treatment of COVID-19 disease or postinfectious conditions is allowed if the last dose of the investigational medicinal product has been received more than 30 days before screening.).
* Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria within the past 60 days prior to initiation of Xultophy® treatment. However, short term insulin treatment for a maximum of 14 days prior to initiation of Xultophy® treatment is allowed, as is prior insulin treatment for gestational diabetes.
* Previous treatment with Xultophy®.
* Female who is known pregnant, breast-feeding or intends to become pregnant.
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.
* Known or suspected hypersensitivity to the active substance or to any of the excipients as specified in the approved Xultophy® label in Japan.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Real-world adult population with type 2 diabetes mellitus in Japan
Sampling Method: Non-Probability Sample
Enrollment: 244 (Actual)
Dates: Start 2021-04-23 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
Change in local laboratory measured HbA1c (Glycated haemoglobin ) | From baseline (Visit 1) to 26 weeks (Visit 3)
  % point

SECONDARY OUTCOMES:
Change in local laboratory measured FPG (Fasting plasma glucose ) | From baseline (Visit 1) to 26 weeks (Visit 3)
  mg/dL
Number of patient-reported non-severe hypoglycaemic after initiation of treatment with Xultophy® | From baseline (Visit 1) to 26 weeks (Visit 3)
  Count of episodes
  Non-severe hypoglycaemia: Defined as an episode with patient reported symptoms and/or self-measured plasma glucose value below 3.9 mmol/L (70 mg/dL). episodes
Number of patient-reported severe hypoglycaemic after initiation of treatment with Xultophy® | From baseline (Visit 1) to 26 weeks (Visit 3)
  Count of episodes
  Severe hypoglycaemia: Defined as an episode of hypoglycaemia requiring assistance of another person to actively administer carbohydrate, glucagon or take other corrective action episodes
Change in concomitant OAD(s) (Oral antidiabetic drugs ) including change in number, class, and frequency of concomitant OAD(s), after initiation of treatment of Xultophy® (Yes/No) | From baseline (Visit 1) to 26 weeks (Visit 3)
  Count of patients
Change in daily dose of Xultophy® | From baseline (Visit 1) to 26 weeks (Visit 3)
  Dose

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (42):
- Japan (42):
  - Seino Internal Medicine Clinic_Internal medicine, Koriyama-shi, Fukushima, Japan
  - Naka Kinen Clinic_Internal medicine, Naka, Ibaraki, Japan
  - Tsuruma Kaneshiro Diabetes Clinic_Internal medicine, Yamato-shi, Kanagawa
  - Jinnouchi Hospital_Internal Medicine, Kumamoto, Kumamoto, Japan
  - Heiwadai Hospital_Internal Medicine, Miyazaki, Miyazaki
  - Abe Diabetes Clinic_Internal Medicine, Ōita, Oita, Japan
  - Asano Clinic, Kawagoe-shi, Saitama, Japan
  - TOSAKI Clinic for Diabetes and Endocrinology_Diabetes and Endocrinology, Aichi
  - Kumanomae Nishimura Naika Clinic_Internal Medicine, Arakawa-ku, Tokyo
  - Yoshida Hospital, Asahikawa-shi, Hokkaido
  - Nippon Medical School Hospital, Diabetes,Metabology,Endocrin, Bunkyo-ku, Tokyo
  - Gengendo Kimitsu Hospital_Diabetes and Endocrinology, Chiba
  - Akaicho Clinic, Chiba-shi, Chiba
  - The Institute of Medical Science, Asahi Life Foundation_Internal Medicine, Chuo-ku, Tokyo
  - Soyokaze CardioVascular Medicine and Diabetes Care, Ehime
  - Futata Tetsuhiro Clinic Meinohama_Internal medicine, Fukuoka-shi, Fukuoka
  - Kawada Clinic, Gunma
  - H.E.C Science Clinic, Kanagawa
  - Chigasaki Municipal Hospital_Endocrinology and Metabolism, Kanagawa
  - Hotaruno hakuyukai Medical Corporation of Japan, Kisarazu-shi, Chiba
  - Gendai Clinic, Kitakyusyu-shi, Fukuoka
  - Ohisama Clinic, Kochi-shi, Kochi
  - Kawasaki Medical School Hospital_Diabetes, Endo and Metabo, Kurashiki-shi, Okayama
  - The Jikei Medical University Hospital_Diabetes, Metabolism and Endo., Minatoku
  - Nakayama Clinic_Nagoya-shi, Aichi, Nagoya-shi, Aichi
  - Abies Kanno Clinic, Numakunai
  - Sumi Clinic, Oita-shi, Oita
  - Oita Endocrinology Diabetes Clinic, Oita-shi, Oita
  - Takagi hospital, Internal Medicine, Okawa-shi, Fukuoka
  - Kansai Electric Power Hospital_Center for Diabetes, Osaka
  - Nakajima Diabetes Clinic, Osaka
  - Matsuda Gastroenterology and Diabetes Clinic, Osaka
  - Okamoto Clinic for Diabetes and Endocrinology, Ōita
  - Budounoki Clinic, Saga-shi, Saga
  - Japan Red Cross Shizuoka Hospital_Diabetes and Endocrinology, Shizuoka
  - Suruga Clinic, Shizuoka-shi, Shizuoka
  - Soka Sugiura Internal Medicine Clinic, Soka-shi, Saitama
  - Higashi Diabetes and Cardiovascular Clinic, Internal, Tamana-shi, Kumamoto
  - Oyama East Clinic_Internal Medicine, Tochigi
  - Clinic Mirai Tachikawa, Tokyo
  - Tamacenter Clinic Mirai, Tokyo
  - Seishinkai Okamoto Naika Iin, Yaizu-shi, Shizuoka

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com